CLINICAL TRIAL: NCT02246322
Title: A Randomized Clinical Trial With a New Needle Device Comparing 25G and 22G Needle in Endoscopic Ultrasound Fine-needle Aspiration of Solid Lesions.
Brief Title: A Clinical Trial With a New Needle Device Comparing Two Needles for EUS_FNA of Solid Lesions.
Acronym: EUS-FNA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Principal Investigator, Michele Tedeschi, MD, Istituto Clinico Humanitas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: BNX-1
Record Dates: First submitted 2014-09-01; First posted 2014-09-22 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2014-09

CONDITIONS: Pancreatic Cancer; Neuroendocrine Tumors; Lymphadenopathies; GIST; Gastric Wall Tumor
Keywords: Pancreatic cancer; Neuroendocrine tumors; Lymphadenopathies; GIST; Gastrointestinal wall neoplasia
MeSH Terms: conditions — Pancreatic Neoplasms; Neuroendocrine Tumors; Lymphadenopathy | interventions — Needles

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 25G needle (Experimental): All consecutive patients that will be referred for solid masses to be aspirated will be randomized to be targeted in the 25G needle arm (A), or in the 22G needle arm (B).
  Interventions: Device: 25G needle
- 22G needle (Experimental): All consecutive patients that will be referred for solid masses to be aspirated will be randomized to be targeted in the 25G needle arm (A), or in the 22G needle arm (B).
  Interventions: Device: 22G needle

INTERVENTIONS:
Device: 25G needle — All consecutive patients that will be referred for solid masses to be aspirated will be randomized to be targeted in the 25G needle arm (A), or in the 22G needle arm (B).
  Arms: 25G needle
Device: 22G needle — All consecutive patients that will be referred for solid masses to be aspirated will be randomized to be targeted in the 25G needle arm (A), or in the 22G needle arm (B).
  Arms: 22G needle

SUMMARY:
Endoscopic ultrasound-guided fine-needle aspiration biopsy (EUS-FNA) is a reliable, safe, and effective technique for obtaining samples from the GI wall lesions and from organs adjacent to the GI tract (pancreas, nodes...).Needles available for EUS-FNA include 25G, 22G and 19G. Some studies have suggested that the 25G needle could be equal or even better than the 22G needle.

The BXN system and neddles are is a newly developed for EUS-FNA. This trial is developed for testing the accuracy of the new neddle system for EUS-FNA and for comparing the two needles types, 25G and 22G.

ELIGIBILITY:
Inclusion Criteria:

* endosonographic appearance of a solid lesions
* age >18 years
* informed consent.

Exclusion Criteria:

* alteration of the coagulation (INR >1.5, PLT <50 x 103 /µL)
* inability to express consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-10 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Clinical performance of 22G and 25G needles | 18 months
  Evaluation of whether enough material for adequate cytological/histological analysis can obtained with equal efficacy with the 25G and the 22G needles. The percentages of adequate samples obtained.

SECONDARY OUTCOMES:
Ease of needle pass | 18 months
  The subjective evaluation of the operator (easy or hard)
Needle malfunction | 18 months
  Needles do not come out of the cover; kinking; needles do not puncture the tissue (presence or absence of malfunction, and registering of the specific malfunction)
Number of passes | 18 months
  The total number of passes needed to obtain adequate material for each lesion (absolute number).
Number of crossovers | 18 months
  The times when the need for passage from the 22G to the 25G needle, or vice versa, registered as percentages of the total procedures.
Major complications | 18 months
  Bleeding (minor: visible at EUS but without clinical significance or less than 2 g/dl; major: dropping of more than 2 g/dl in Hb levels and clinically significant), perforation (presence/absence), infection (need for hospitalization).

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Carrara, MD, Principal Investigator — Humanitas Research Hospital IRCCS, Rozzano-Milan
Locations (1):
- Humanitas Research Hospital, Rozzano, Milan, Italy

REFERENCES:
- [Background] Camellini L, Carlinfante G, Azzolini F, Iori V, Cavina M, Sereni G, Decembrino F, Gallo C, Tamagnini I, Valli R, Piana S, Campari C, Gardini G, Sassatelli R. A randomized clinical trial comparing 22G and 25G needles in endoscopic ultrasound-guided fine-needle aspiration of solid lesions. Endoscopy. 2011 Aug;43(8):709-15. doi: 10.1055/s-0030-1256482. Epub 2011 May 24. PMID 21611946
- [Background] Siddiqui UD, Rossi F, Rosenthal LS, Padda MS, Murali-Dharan V, Aslanian HR. EUS-guided FNA of solid pancreatic masses: a prospective, randomized trial comparing 22-gauge and 25-gauge needles. Gastrointest Endosc. 2009 Dec;70(6):1093-7. doi: 10.1016/j.gie.2009.05.037. Epub 2009 Jul 28. PMID 19640524